CLINICAL TRIAL: NCT03802708
Title: Fetal Alcohol Spectrum Disorder-Is This a Ciliopathy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Helly Goez, Principal Investigator, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00076905
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Fetal Alcohol Spectrum Disorder
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Intervention Model Description: pilot. 5 children with FASD- 5 healthy children
Masking Description: this is N/A
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- control (Other): control
  Interventions: Diagnostic Test: Metabolomic analysis urine sample

INTERVENTIONS:
Diagnostic Test: Metabolomic analysis urine sample — a urine sample will be anlayzed for metabolic pathways involving Nitric Oxide Nitric Oxide level will be measured at the exhaled air sample
  Other Names: NO- Analyzer breath test

SUMMARY:
Urine sample and exhaled Nitric Oxide will analyzed and compared between children diagnosed with Fetal Alcohol Spectrum Disorder and healthy control.

Pilot study- 5 children in each group

DETAILED DESCRIPTION:
Background: The term "fetal alcohol spectrum disorder" (FASD) describes a broad spectrum of neurodevelopmental presentations resulting from alcohol exposure in utero. The prevalence has been estimated at 1 in 100 people, and estimated to be more than 330 000 affected individuals in Canada. The Canadian Diagnostic Guidelines describe the physical and neurodevelopmental effects resulting from prenatal alcohol exposure. These include distinct facial features, microcephaly and neurodevelopmental deficits.

Ethanol toxicity is researched in association to the concentration, duration, and timing of ethanol exposure and the possible pathways leading to phenotypic translation to teratogenesis. Studies of FASD in animal models are beginning to implicate a number of susceptibility genes that are involved in various molecular pathways on gene-ethanol interactions. Some of which are reportedly involved in ethanol teratogenesis as a part of their roles in DNA damage control, Central Nervous System axis formation, cellular survival as well as proliferation and growth.

A mutation in one particular gene, neuronal nitric oxide synthase (nNOS)) is known to worsen alcohol induced neuronal death both in vivo and in vitro, and expression of the nNOS gene protects neurons against alcohol toxicity Nitric Oxide (NO) is synthesized by the enzyme nitric oxide synthase (NOS through) L-arginine There are three NOS isoforms: neuronal NOS (nNOS, NOS-1), inducible NOS (iNOS, NOS-2), and endothelial NOS (eNOS, NOS-3) .NO is associated with modulation of neurotransmission and memory formation along with other vital activities. In the presence of O2, radicals form that can lead to toxicity. They may be disruptive to cell signaling processes and result in pathological conditions.

Data suggest that ethanol alters NOS expression and activity in the brain There are known effects of ethanol on production of NO, NOS activities, and interactions of NO with alcohol metabolism enzymes.

Dose and length of ethanol exposure are the main factors determining ethanol effects on NO production, NOS activity or NOS expression.

Structural congenital brain anomalies are described in the context of FASD including microcephaly, migration anomalies, neural tube defects along with midline brain anomalies involving the corpus callosum, cerebellar anomalies and hydrocephalus.

Cilia are evolutionarily-conserved antennae-like organelles found on the surface of cells. Cilia detect different extracellular stimuli such as fluid flow, light, smell, and hormones through specific ciliary receptors, and they play key roles in cell locomotion and division, fluid movement, as well as embryonic development of different tissues. In regards to neural development, ciliary growth factors were recently shown to play a role in embryonic neuronal cell migration and signaling as well as in formation of the Central Nervous System (CNS) midline and lateralization. In the mature organism, cilia extend from the basal bodies of the ependymal cells lining the ventricular surface of the brain, where they facilitate the flow of Cerebro Spinal Fluid (CSF).

Nervous system defects are strongly associated with a number of ciliopathies, with common findings including midline defects such as hydrocephalus, neural tube defects, and a plethora of cortical and cerebellar abnormalities.

The prototype human ciliary disease has been Primary Ciliary Dyskinesia (PCD). In the past decade, significant advancement in understanding of PCD has led to improved diagnosis, mainly by the finding that Nasal nitric oxide (nasal NO) is greatly reduced in these patients. The mechanism of this reduction has been suggested to be related to reduced iNOs expression as part of the ciliopathy. Nasal NO measurement is a simple non-invasive test easily carried out even in the youngest patients.

As NO measurement is a simple non-invasive test with immediate results, it serves as an ideal screening test for suggestive diagnosis of various ciliopathies, including those involving brain malformations.

In recent work, this research group was the first to determine a connection between ciliary dysfunction as measured by nasal NO concentration and isolated midline central nervous system (CNS) anomalies The overall mean nasal NO level in children with isolated midline CNS anomalies in the study, was significantly lower compared to the previously-established normal range with some being within the range of Primary Ciliary Dyskinesia (PCD). Recent work shows that inter neuronal connectivity, brain ventricles morphogenesis and proper formation of the neural tube depend on non-disrupted ciliary function.

The primary cilia function as a result of membrane proteins such as polycystin-1 (PC-1), PC-2, TRPV4, P2Y12, and fibrocystin. Acetylated alpha tubulin is a known ciliary marker.

Alterations in PC-1 are associated with polycystic kidney disease type 1 mutations that were found to be associated with fatty acid oxidation defects in metabolomic and lipidomic tests. Acetylated alpha tubulin is assessed through proteinomic analysis.

Hypothesis: Given the recent recognition of the interactions between NO with ethanol and the important role of cilia in early brain development, the investigators hypothesize that cilia may be involved in molecular pathways leading to brain injury in children that are diagnosed with FASD. Such a mechanism has not been previously explored.

The investigators hypothesize that nasal NO levels as well as the key metabolites in patients diagnosed with FASD will be reduced compared to healthy controls.

Objective: This study will aim at measuring nasal NO in a selected group of patients diagnosed with Fetal Alcohol Spectrum Disorder, along with metabolomics and proteinomic analysis as related to key metabolites involved in NO pathway in urine samples, and compare them to healthy children. This study will enable clinicians to potentially employ a non-invasive screening tool for pediatric patients with suspected Fetal Alcohol Spectrum Disorder and consider an early developmental intervention.

Methods: 10 children ages 5-16 years, who are diagnosed with FASD will be recruited from the FASD outpatient clinic at the Glenrose Rehabilitation Hospital. 10 healthy children of the same age range will be recruited through the HICUPP registry for healthy children (Pro00056156).

The investigators will measure nasal NO levels by inserting an inert NO sampling line with a disposable foam olive (DirectMed Inc., Glen Cove, NY) into the child's nostril while the contralateral nostril is left open. Air will be then sampled at a constant rate of 0.3 liters/min from the nose by a chemiluminescent analyzer which provides measurement of the nasal NO level in parts per billion (ppb). All nasal NO measurements will be performed with the subjects seated.

Measurements will be obtained using an NO analyzer (CLD 88 SP, ECO PHYSICS AG, Duerten, Switzerland). The analyzer will be calibrated according to the manufacturer's specifications. Measurements will be made using velum-closure technique via exhalation from a deep inspiration through a fixed resistor (disposable, cardboard cylinder with 1 mm opening; DirectMed Inc., Glen Cove, NY) for 20-40 seconds or via a party favor blowout toy with a comparable expiratory resistance. Both types of resistor require slight puffing of the cheeks to develop a mouth pressure > 5 cm H2O, a pressure sufficient to close the soft palate. The maneuvers will be performed according to ATS/ERS guidelines. In patients who are uncooperative with the above maneuver the measurements will be made using tidal breath sampling.

The examiner will enter the measured NO level directly into a computer file, which will be saved in an encrypted format on a password-protected computer at the Glenrose Rehabilitation Hospital. Identifying information such as participants' names or phone numbers will not be entered. Each participant will be assigned a number instead of a name, which will be recorded. Other identifying information, such as the child's gender, age and diagnosis, will be coded using a number as well.

Based on information provided, a statistical analysis of co-variants will be performed, comparing the measured NO levels of patients with FASD to healthy controls (with the reference range of the normal as published in Mateo 2011 and Marthin 2011).

In addition to the nasal NO measurements, the investigators will also conduct metabolomic and proteomic analysis to measure the levels of key metabolites and proteins in urine of patients with FASD. These will be compared to the healthy, controls to further explore this hypothesis of ciliary involvement. The metabolomic analyses will be used to measure key metabolites involved in the NO pathway (arginine, citrulline, ornithine, asymmetric dimethylarginine) as well as soluble NO byproducts (nitrotyrosine, nitrotryptophan, and 3-nitro-4-hydroxyphenylacetic acid). Additional metabolomic studies will be performed to look for altered beta-oxidation markers (acylcarnitines) which can be affected by ciliary dysfunction, vitamin levels (esp. vitamin A and its byproducts) as well as changes in catecholamines (due to altered neuronal functions affected by cilia) in urine. The metabolomic analyses will be done using targeted, MS-based metabolomics methods. The investigators will also conduct proteomic analysis on urine in FASD patients to measure changes in key ciliary proteins, namely polycystin-1 (PC-1)( PC-2, TRPV4, P2Y12, fibrocystin) as well as acetylated alpha-tubulin and compare these values to a group of healthy children. The proteomic analyses will consist of a combination of MS-based proteomics and immunoassays.

Data will be analyzed using PASW Statistics Version 19 (SPSS Inc., 2010). Alpha will be set at .05 for all analyses. The percentage of children who score above and below age and norm-based cut-off values on each measurement will be computed.

To determine whether the two groups (FASD, Healthy controls) differ in the measured level a Multivariate Analysis of Variance (MANOVA) will be conducted on subscale scores using Group as a between-subjects factor.

Noting that the sample size is small, the investigators will report an effect size between the groups for the NO level, and the metabolomics analysis, as well as a 95% confidence interval for the effect size. The hypothesis is that there is a difference between the groups; given that the investigators cannot prove the null (i.e., a lack of a statistically significant finding will not prove the hypothesis), the investigators will use this effect size to instead estimate the effect. However it is hypothesized that the nasal NO levels and key metabolites as relates to NO in children with FASD will be reduced in comparison to healthy controls.

Following the completion of the study, the de-identified data will be kept in an encrypted file on the password-protected computer for a minimum of five years.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 5-16
* Diagnosis of FASD

Exclusion Criteria:

* Sinopulmonary anomaly
* Cardiac anomaly
* Asthma
* Previously known Genetic condition
* Previously known Metabolic condition
* Polypharmacy

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Nitric Oxide metabolites in urine | At time of enrollment
  metabolomic analysis

SECONDARY OUTCOMES:
nitric oxide concentration | At time of enrollment
  NO-Analyzer breath test

CONTACTS AND LOCATIONS:
Locations (1):
- Glenrose rehabilitation hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
results from analysis will be available